CLINICAL TRIAL: NCT01977300
Title: Atypical Antipsychotics for Continuation and Maintenance Treatment After an Acute Manic Episode
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Eli Lilly and Company (Industry); Janssen-Ortho Inc., Canada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H02-70188; V02-0130 (Other: Vancouver Coastal Health Research Institute)
Record Dates: First submitted 2013-10-22; First posted 2013-11-06 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2013-10

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — Valproic Acid; Lithium; Lithium Carbonate; Risperidone; Olanzapine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mood stabilizer & Placebo (Placebo Comparator): Patients will receive lithium or valproate plus placebo for 52 weeks (risperidone or olanzapine tapering will begin on the day of randomization with discontinuation of the drug within 2 weeks).
  Interventions: Drug: Valproate; Drug: Lithium; Other: Placebo
- '24 week " arm (Experimental): Continuation of the lithium or valproate plus risperidone or olanzapine for 24 weeks followed by mood stabilizer plus placebo for another 28 weeks. Dosages: 1 to 6 mg of risperidone, 5 to 20 mg olanzapine.
  Interventions: Drug: Valproate; Drug: Lithium; Drug: Risperidone; Drug: Olanzapine; Other: Placebo
- "52 week" arm (Active Comparator): Continuation of the atypical antipsychotic, risperidone or olanzapine, plus lithium or valproate for 52 weeks.
  Interventions: Drug: Valproate; Drug: Lithium; Drug: Risperidone; Drug: Olanzapine

INTERVENTIONS:
Drug: Valproate — serum level of 50 to 125 ug/L
  Other Names: Valproic Acid
Drug: Lithium — serum levels of 0.6 to 1.2 mmol/L
  Other Names: Lithium Carbonate
Drug: Risperidone — 1 to 6 mg/day
  Other Names: Risperdal
  Arms: "52 week" arm; '24 week " arm
Drug: Olanzapine — 5 to 25 mg/day
  Other Names: Zyprexa
  Arms: "52 week" arm; '24 week " arm
Other: Placebo — manufactured to mimic risperidone and olanzapine
  Other Names: Sugar Pill
  Arms: '24 week " arm; Mood stabilizer & Placebo

SUMMARY:
Hypothesis: Continuation of an atypical antipsychotic medication in combination with a Mood Stabilizer, following remission from an acute manic episode, lowers the rates of relapse and recurrence of mood episodes compared to discontinuing the antipsychotics within days of resolution of manic symptoms.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo controlled trial over 52 weeks. Patients will be on one of four combinations of medications at the time of entry into the study: a) lithium and risperidone, b) lithium and olanzapine, c) valproate and risperidone, or d) valproate and olanzapine. After obtaining informed consent, patients will be randomised to one of three groups 1)"0" week group: patients will receive lithium or valproate plus placebo for 52 weeks (risperidone or olanzapine tapering will begin on the day of randomisation with discontinuation of the drug within 2 weeks), 2) continuation of the same atypical antipsychotic, risperidone or olanzapine, plus lithium or valproate for 24 weeks (tapering of the antipsychotic begins at the end of 24 weeks and completed within 2 weeks) followed by the same mood stabilizer plus placebo for another 28 weeks, and 3) continuation of the atypical antipsychotic, risperidone or olanzapine, plus lithium or valproate for 52 weeks. The duration of the double-blind phase of the study will be 52 weeks and all patients will continue on the mood stabilizer, lithium or valproate, they had been on during the acute mania for the full duration of the study. The serum level of the mood stabilizer will be maintained within the therapeutic range (0.6 to 1.2 mmol/L for lithium and 50 to 125 ug/L for valproate) throughout the 52 weeks as determined by blood tests. The dose and the type of atypical antipsychotic (ie risperidone or olanzapine) each patient will receive during the double-blind period will be the same that the patient had been on at the time of entry into the double-blind phase. All patients, irrespective of which treatment arm they are in, will receive active psychoeducation and counselling regarding sleep hygiene, healthy daily routines and rhythms, alcohol and substance abuse, anxiety management, conflict resolution and problem solving as clinically indicated in routine clinical practice. Patients who withdraw from or meet a primary end point of the study will be treated actively as done in regular clinical practice.

Patients will not be allowed to receive any other psychotropic medication with the exception of benzodiazepines for sedation and anti-parkinsonian medication for extrapyramidal side effects. The doses of these will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were recently (within the last 12 weeks) commenced on treatment for a Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) manic or mixed episode with a combination of lithium and risperidone, lithium and olanzapine, valproate and risperidone, or valproate and olanzapine;
* Patients on 1 to 6 mg of risperidone or 5 to 25 mg of olanzapine
* Patients who are in remission from mania for at least 2 weeks but no more than 6 weeks and have maintained remission for 2 consecutive weeks;
* Patients must not be taking any other psychotropic medication (with the exception of benzodiazepines) or treatments including bromocriptine, omega 3 fatty acids, Axid or EMPower;
* Patients aged 17 and above.

Exclusion Criteria:

* Any subjects who do not meet the above inclusion criteria will be excluded from the study.
* In order for the findings to be generalizable to clinically representative patients with bipolar disorder, any patients with a history of co-morbid substance abuse or medical illnesses will not be excluded.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2003-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the time to any mood episode (depressive or manic episode). | 52 weeks
  A mood episode is defined as 1) Young Mania Rating Scale (YMRS) score of 15 or greater 2)Hamilton Rating Scale for Depression (HAM-D) 21-item score of 15 or greater or a HAM-D suicide item score of 3 or greater 3)A Clinical Global Impression -Severity (CGI-S) score of 3 or greater 4) a patient requiring hospitalization for treatment of mood symptoms or 5) a patient who makes a suicide attempt or commits suicide during the study.

SECONDARY OUTCOMES:
Time to manic episode. | 52 weeks
  Time to occurrence of a manic episode measured by Young Mania Rating Scale (YMRS) score of 15 or greater .
Time to depressive episode | 52 weeks
  Time to occurrence of a depressive episode measured by Hamilton Rating Scale for Depression (HAM-D) 21-item score of 15 or greater or a HAM-D suicide item score of 3 or greater.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi N Yatham, Dr., Principal Investigator — University of British Columbia; Serge Beaulieu, Dr., Study Director — McGill University, Montreal; Andree Daigneault, Dr., Study Director — Clinique des Maladies Affectives, Montreal; Verinder Sharma, Dr., Study Director — Regional Mental Health Care London, Ont.; Hubert Wong, Dr., Study Director — University of British Columbia; Ayal Schaffer, Dr., Study Director — Sunnybrook Health Sciences Centre, Toronto, Ont.; Sagar Parikh, Dr., Study Director — Centre for Addiction and Mental Health, Toronto, Ont.; Philippe Baruch, Dr., Study Director — Clinique des troubles de l'humeur, Quebec; Peter Silverstone, Dr., Study Director — University of Alberta; Roumen Milev, Dr., Study Director — Providence Continuing Care, Kingston, Ont.; Ram Veluri, Dr., Study Director — Northern Health Research Inc., Sudbury, Ont.; Pablo Cervantes, Dr., Study Director — Montreal General, Quebec; Claire O'Donovan, Dr., Study Director — Mental Health Services, Halifax, NS; Flavio Kapczinski, Dr., Study Director — Hospital de Clinicas de Porto Alegre, Porto Alegre, Brazil; Benny Lafer, Dr., Study Director — Instituto de Psiquiatria do Hospital das Clínicas, Sao Paulo, Brazil; Angelo B Miralha da Cunha, Dr., Study Director — Santa Maria, Brazil; Joao Quevedo, Dr., Study Director — Casa de Saude do Rio Maina Ltda, Criciuma, Brazil
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Yatham LN, Beaulieu S, Schaffer A, Kauer-Sant'Anna M, Kapczinski F, Lafer B, Sharma V, Parikh SV, Daigneault A, Qian H, Bond DJ, Silverstone PH, Walji N, Milev R, Baruch P, da Cunha A, Quevedo J, Dias R, Kunz M, Young LT, Lam RW, Wong H. Optimal duration of risperidone or olanzapine adjunctive therapy to mood stabilizer following remission of a manic episode: A CANMAT randomized double-blind trial. Mol Psychiatry. 2016 Aug;21(8):1050-6. doi: 10.1038/mp.2015.158. Epub 2015 Oct 13. PMID 26460229